CLINICAL TRIAL: NCT02280564
Title: Pilot Study of A Cell-Phone System to Improve Health of Youth With Diabetes
Brief Title: Study of A Cell-Phone System to Improve Health of Youth With Diabetes
Acronym: FL3X
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Elizabeth Mayer-Davis, PhD, Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-0240; R21DK085483-01 (NIH)
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Type 1 Diabetes
Keywords: motivational interviewing; problem solving skills; family communication; technology support; cell phone system
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Standard diabetes care
- Health coaching with technology support (Experimental): Behavioral strategies including problem solving skills building, family communication counseling, technology support, motivational interviewing support.
  Interventions: Behavioral: health coaching with technology support

INTERVENTIONS:
Behavioral: health coaching with technology support — Intensive behavior change support. Engaging participants to take an active role in their diabetes care using motivational interviewing, technology, family communication, problem solving skills.
  Other Names: FL3X
  Arms: Health coaching with technology support

SUMMARY:
FL3X is an integrated diabetes self-management system that incorporates modern cell phone technology with behavioral modification approaches to improve diabetes self-management in high-risk youth. Utilizing such approaches will increase adherence to diabetes management behaviors and improve glucose control by providing increased autonomy over diabetes care.

DETAILED DESCRIPTION:
FL3X utilizes diabetes care providers (diabetes educators) as health coaches to employ behavioral modification techniques including motivational interviewing and problem solving skills training. Coaches help adolescents and their families learn these techniques to improve diabetes self management behaviors and diabetes care.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes with duration at least 12 months
* between ages 12-16 years at registration
* poor glycemic control (A1c 8.0-13.0%)
* parent/guardian willing to also participate
* minority race/ethnicity
* low income

Exclusion Criteria:

* pregnant (if female)
* diabetes type 2 or gestational
* no health insurance
* Pre-existing systemic chronic disease (drug abuse, cancer, psychiatric conditions)

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2011-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in HbA1c at 4 months | 4 months

SECONDARY OUTCOMES:
Change from Baseline in Quality of Life measures at 4 months | 4 months
  Quality of Life will be assessed via self report questionnaire data.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Mayer-Davis, PhD, Principal Investigator — UNC-CH
Locations (3):
- United States (3):
  - University of Colorado Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - WakeMed Hospital, Raleigh, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio